CLINICAL TRIAL: NCT05290038
Title: ARON-2 Study-Multicentric International Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Matteo Santoni (Other)
Responsible Party: Sponsor-Investigator, Matteo Santoni, Oncologist, Hospital of Macerata
Organization: Hospital of Macerata (Other)
Other Study IDs: ARON-2
Record Dates: First submitted 2022-02-22; First posted 2022-03-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
Keywords: immunotherapy; real world experience; efficacy of pembrolizumab; artificial intelligence technology; Artificial Neural Network
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The ARON-2 study retrospectively analyze patients treated with pembrolizumab as first-line therapy in patients platinum-unfit or as second-line therapy in patients progressed after previous platinum-based chemotherapy. The amendment has been designed to also analyze patients treated with enfortumab vedotin progressed to previous platinum-based chemotherapy and anti-PD-1/PD-L1 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18y
* Histologically confirmed diagnosis of UC of upper and/or lower urinary tract
* Histologically or radiologically confirmed metastatic disease
* Patients treated with at least one of the following:
* Treatment with pembrolizumab in patients progressed after previous platinum-based chemotherapy or as first-line therapy in patients platinum-unfit, and at least 1 cycle of pembrolizumab within the period from 1 January 2018 to 30 November 2021
* Treatment with enfortumab vedotin in patients progressed to previous platinum-based chemotherapy and anti-PD-1/PD-L1 inhibitor and at least 1 cycle of enfortumab vedotin within the period from June 1st 2022 to July 31st 2023

Exclusion Criteria:

* Patients without histologically confirmed diagnosis of UC
* Patients without histologically or radiologically confirmed metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with pembrolizumab as first-line therapy in patients platinum-unfit or as second-line therapy in patients progressed after previous platinum-based chemotherapy, or patient treated with enfortumab vedotin progressed to previous platinum-based chemotherapy and anti-PD-1/PD-L1 inhibitor.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) of patients with metastatic Urothelial Cancer (UC) treated with pembrolizumab or enfortumab vedotin | November 15th, 2023
Progression-Free Survival (PFS) of patients with metastatic Urothelial Cancer (UC) treated with pembrolizumab or enfortumab vedotin | November 15th, 2023
Overall Response Rate (ORR) of patients with metastatic Urothelial Cancer (UC) treated with pembrolizumab or enfortumab vedotin | November 15th, 2023

SECONDARY OUTCOMES:
prognostic role of smoking attitude, obesity and concomitant medications in patients treated with pembrolizumab or enfortumab vedotin | November 15th, 2023
  Statistical analysis of data obtained by medical charts related to smoking attitude, obesity and concomitant medications in patients with metastatic UC treated with pembrolizumab or enfortumab vedotin

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Macerata, UOC Oncologia, Macerata, Macerata, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzo M, Morelli F, Urun Y, Buti S, Park SH, Bourlon MT, Grande E, Massari F, Landmesser J, Poprach A, Takeshita H, Roviello G, Myint ZW, Popovic L, Soares A, Abahssain H, Giannatempo P, Molina-Cerrillo J, Incorvaia L, Salah S, Zeppellini A, Monteiro FSM, Porta C, Gupta S, Santoni M. Real-Life Impact of Enfortumab Vedotin or Chemotherapy in the Sequential Treatment of Advanced Urothelial Carcinoma: The ARON-2 Retrospective Experience. Cancer Med. 2025 Feb;14(4):e70479. doi: 10.1002/cam4.70479. PMID 39980145